CLINICAL TRIAL: NCT05407649
Title: Abscopal Effect and Safety of Recurrent and Refractory Advanced Thymic Epithelial Tumours Treated With Combined Therapy of Local Radiotherapy and Granulocyte-macrophage Colony-stimulating Factor
Brief Title: Abscopal Effect of Radiotherapy in Combination With rhGM-CSF for Advanced Thymic Epithelial Tumours
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Cancer Hospital, China (Other)
Responsible Party: Principal Investigator, Fan Min, Clinical Professor, Shanghai Cancer Hospital, China
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUSCC-SGCI001
Record Dates: First submitted 2022-05-30; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Thymoma
MeSH Terms: conditions — Thymoma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy Combined with GM-CSF (Experimental)
  Interventions: Radiation: Radiotherapy Combined with GM-CSF

INTERVENTIONS:
Radiation: Radiotherapy Combined with GM-CSF — Patients with stable or progressing metastatic thymic epithelial tumours, with at least two distinct measurable sites of disease, were treated with concurrent radiotherapy (35 Gy in ten fractions or 60Gy in 30 fractions) to one metastatic site and granulocyte-macrophage colony-stimulating factor (125 μg/m(2) subcutaneously injected daily for 2 weeks, starting during the second week of radiotherapy).

SUMMARY:
The purpose of this study is to determine whether radiotherapy (RT) combined with recombined human granulocyte-macrophage colony stimulating factor(rhGM-CSF) is safe, effective in the treatment of patients with advanced thymic epithelial tumours.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Histologically proven thymic epithelial tumours；
3. Stage IV according to UICC stage system(version 8,2017), at least with two evaluable abscopal lesions (≥1cm)（excluding intestinal metastasis）;
4. Evaluated as effective or stable disease after first-line chemotherapy or progressed after second-line chemotherapy (progression sites were no more than three sites);
5. ECOG performance status: 0-1;
6. Life expectancy ≥ 3 months.
7. Adequate baseline organ and marrow function: absolute neutrophil count greater than 1500 cells per μL, platelet concentration of greater than 50 000 per μL, total bilirubin less than 1•5 times the upper limit of normal (ULN), aspartate aminotransferase and alanine aminotransferase less than 2•5 times the ULN, and serum creatinine less than 1•5 times the ULN;
8. Female subjects have a negative urine or serum pregnancy test within 1 week prior to treatment if of childbearing potential;
9. Asymptomatic subjects with brain metastasis can be included, but the sites of brain cannot be considered as target sites;
10. Asymptomatic subjects with bone metastasis can be included, but the sites of bone cannot be considered as target sites.

Exclusion Criteria:

1. Having received immunotherapy within 4 weeks prior to inclusion;
2. Allergic to GM-CSF, INF-α2b or diagnosed with immune system disease, receiving immunosuppressant, such as prednisone, dexamethasone, methylprednisolone, methotrexate, hydroxychloroquine, cyclophosphamide, azathioprine and so one;
3. Receiving treatment of other trials;
4. Any unstable systemic disease, including active infection, symptomatic congestive heart failure,myocardial infarction onset six months before included into the group, unstable angina, and severe arrhythmia, uncontrolled chronic lung disease;
5. Unwilling to sign consent;
6. Women in pregnancy or lactation;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
The abscopal effect rate | up to 12 months
  The proportion of patients with an abscopal response assessed after the initiation of treatment
  The proportion of patients with an abscopal response assessed after the initiation of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No